CLINICAL TRIAL: NCT03325530
Title: A Collaborative Approach to Providing Healthy Food Access and Sustainable Physical Activity Opportunities at Boy Scouts of America Summer Camp
Brief Title: Providing Healthy Food Access and Physical Activity Opportunities at Boy Scouts of America Summer Camp
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Boy Scouts of America (Unknown)
Responsible Party: Principal Investigator, Jennifer Kraschnewski, Associate Professor of Medicine, Pediatrics, and Public Health Sciences Executive Director, Penn State PRO Wellness Associate Director of Research, Division of General Internal Medicine, Milton S. Hershey Medical Center
Other Study IDs: STUDY00005462
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Childhood Obesity
Keywords: Adolescent; Nutrition; Physical Activity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focus Group
  Interventions: Behavioral: Focus Group with Participants

INTERVENTIONS:
Behavioral: Focus Group with Participants — Focus groups with leaders (18+) to investigate tolerance to healthy initiatives

SUMMARY:
To measure impact of improved healthy food access and physical activity opportunities at summer Boy Scout camp, a four-week intervention to address nutrition and physical activity with youth (n=911) and adults (n=247) was conducted at Bashore Scout Reservation in Jonestown, Pennsylvania between June and July of 2016. Intervention components included dining hall menu modifications, healthy messaging, introduction of nutritious snacks available for purchase, and a physical activity challenge.

Menu modifications resulted in improved satisfaction scores related to portion sizes (+28%) and variety (+14%), decreased plate waste, and consistent food costs. Introduction of nutritious snacks at Trading Post resulted in increased satisfaction (+13%) and increased sales per person (+20%). Physical activity increased (+22%) as a result of a step competition between troops. Small changes towards a healthier camp were widely accepted and successful, indicating potential for translation to other camps within the organization.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years
2. Sex: Male or female
3. Fluent in written and spoken English
4. Boy Scout staff, troop leader or parent of Boy Scout camper

Exclusion Criteria:

1. Not Fluent in written and spoken English
2. Non Boy Scout stafftroop leader or not a parent of a Boy Scout camper
3. Decisional impairment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Boy Scout staff, troop leader or parent of Boy Scout camper
Sampling Method: Non-Probability Sample
Enrollment: 1158 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of intervention as assessed through focus groups and evaluation surveys | June 2016- August 2016
  Feedback from troop leaders informed researchers concerning how scouts felt about and how receptive scouts are to healthy initiatives.

IPD SHARING:
Plan to Share IPD: No